CLINICAL TRIAL: NCT04682184
Title: A Study to Investigate Continuous Heart Rate Monitoring Using a Chest-worn Biosensor on the Background of Drug-induced Positive and Negative Heart Rate Changes
Brief Title: A Study of Continuous Heart Rate Monitoring in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18168; H6O-MC-O016 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-10; First posted 2020-12-23 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Propranolol; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wearable Biosensor Patch Device + Propranolol (Experimental): Participants will wear the biosensor patch device followed by propranolol administered orally in one of three study periods.
  Interventions: Drug: Propranolol; Device: Wearable Biosensor Patch Device
- Wearable Biosensor Patch Device + Pseudoephedrine (Experimental): Participants will wear the biosensor patch device followed by pseudoephedrine administered orally in one of three study periods.
  Interventions: Drug: Pseudoephedrine; Device: Wearable Biosensor Patch Device
- Wearable Biosensor Patch Device (Alone) (Experimental): Participants will wear biosensor patch device (alone) during one of three study periods.
  Interventions: Device: Wearable Biosensor Patch Device

INTERVENTIONS:
Drug: Propranolol — Administered orally.
  Arms: Wearable Biosensor Patch Device + Propranolol
Drug: Pseudoephedrine — Administered orally.
  Arms: Wearable Biosensor Patch Device + Pseudoephedrine
Device: Wearable Biosensor Patch Device — Biosensor patch device attached to the chest and worn throughout the trial with replacement of biosensor every 7 days.

SUMMARY:
The main purpose of this study in healthy participants is to find out whether a heart rate monitor will accurately pick up changes in heart rate caused by 2 different medications (pseudoephedrine and metoprolol), on the background of daily activities. Participants will wear a patch heart rate and activity monitor on the chest for the entire study. The study will last about 36 days and may include up to seven visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Have a body mass index (BMI) of 18.0 to 35 kilograms/square meter (kg/m2), inclusive at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have history of sensitive skin or chronic skin conditions, like eczema
* Regularly use known drugs of abuse
* Are women who are pregnant or lactating
* Have known allergies to medications used in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
The mean change in heart rate (HR) | Day 1: Hour 1, Hour 4 post intervention
  The mean change in HR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No